CLINICAL TRIAL: NCT03541252
Title: Tolerability of Laser-assisted Cisplatin + 5-fluorouracil- an Exploratory Proof of Concept Study of Topical Combination Chemotherapy for Basal Cell Carcinoma
Brief Title: Topical Laser-assisted Combination Chemotherapy for Basal Cell Carcinoma- a Clinical Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merete Haedersdal (Other)
Responsible Party: Sponsor-Investigator, Merete Haedersdal, Professor, Senior Consultant, PhD, DMSc, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT2018-000141-39
Record Dates: First submitted 2018-04-25; First posted 2018-05-30 (Actual); Results first posted 2022-03-15 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-03

CONDITIONS: Carcinoma, Basal Cell
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Intervention Model Description: A prospective clinical, uncontrolled, open-label, explorative phase IIa trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Basal Cell Carcinoma Patients (Experimental): Patients (>18 years) with histologically-verified superficial or nodular basal cell carcinoma (<20 mm on the face/scalp, <50mm on the trunk/extremities)
  Interventions: Drug: AFL-assisted cisplatin+5-FU

INTERVENTIONS:
Drug: AFL-assisted cisplatin+5-FU — Patients will receive AFL-assisted cisplatin+5-FU as a treatment for their BCC. In brief, treatment areas consisting of tumors and a 5 mm margin will undergo CO2 laser exposure followed by 60 min topical application of a marketed and commercially available IV cisplatin solution (0.1%) After removal of cisplatin, a commercially distributed 5-FU cream (5%) will be applied to the treatment area at a dose of 0.125 ml per cm2 and left under occlusion. After skin evaluations on Day 1 and 5 after treatment, the same 5-FU dose will be applied, again left under occlusion. In total, 5-FU will remain on the skin for 7 days after AFL treatment whereafter it will be washed off. An additional repeat AFL-cisplatin+5-FU treatment on Day 30 will be offered if tumors persist, based on clinical evaluation and imaging on Day 30.

SUMMARY:
A prospective clinical, uncontrolled, open-label, explorative phase IIa trial on patients with histologically- confirmed superficial and nodular basal cell carcinoma (BCC) . The study assesses tolerability and tumor clearance after laser-assisted topical delivery of two synergistic chemotherapeutic agents, cisplatin and 5-fluorouracil (5-FU) in BCC patients.

DETAILED DESCRIPTION:
Patients will receive ablative fractional laser (AFL)-assisted cisplatin+5-fluorouracil (5-FU) as a treatment for their cutaneous basal cell carcinoma (BCC). In brief, treatment areas consisting of tumors and a 5 mm margin will undergo AFL exposure (CO2 laser) followed by 60 min topical application of a marketed and commercially available IV cisplatin solution (0.1%) at a dose of 0.25 ml per cm2. After removal of cisplatin, a commercially distributed 5-FU cream (5% Efudix®) will be applied to the treatment area at a dose of 0.125 ml per cm2 and left under occlusion. After skin evaluations on Day 1 and 5 after treatment, the same 5-FU dose will be applied, again left under occlusion. In total, 5-FU will remain on the skin for 7 days after AFL treatment whereafter it will be washed off.

An additional repeat AFL-cisplatin+5-FU treatment on Day 30 will be offered if tumors persist, based on clinical evaluation and imaging on Day 30.

Outcome measures and methods/techniques are summarized below.

Primary outcome:

To investigate tolerability of topical AFL-assisted cisplatin+5-FU therapy for BCC by evaluating:

I. Severity and duration of clinical local skin reactions including erythema, edema, scabbing, flaking and pustulation assessed by a physician using an established 0-4 point scale (none, mild, moderate, severe) from 0-30 days post-treatment.

II. Occurrence of side effects (prolonged erythema/edema, hyper/hypopigmentation, scarring and infection) up to 3 months post-treatment.

Secondary outcome:

1) To monitor BCC tumor size and clearance based on clinical assessments and dermoscopy, supported by non-invasive imaging techniques including dynamic optical coherence tomography (D-OCT), reflectance confocal microscopy (RCM), high intensity focused ultrasound (HIFU) and histological analysis up to 3 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-verified, previously untreated superficial or nodular BCCs on the scalp, face, extremities or trunk
2. >18 years of age at baseline
3. Legally competent, able to give verbal and written informed consent
4. Subject in good general health, is willing to participate and can comply with protocol requirements.
5. Fitzpatrick skin phototype I-III
6. Female subjects of childbearing potential1 must be confirmed not pregnant by a negative urine pregnancy test prior to trial treatment.

Exclusion Criteria:

1. High-risk BCC i. Tumors in the following anatomical locations: midface, orbital, ears ii. Size: >20 mm in facial/scalp areas or > 50 mm in non-facial/non-scalp areas iii. Subtype: morpheaform and micronodular BCC iv. History: Gorlin syndrome or immunosuppression
2. Previous treatment of the BCC lesion
3. Known allergy to cisplatin or Efudix®
4. Other skin diseases present in the treatment area
5. Tattoo in the treatment area which may interfere with or confound evaluation of the study
6. History of keloids which is deemed clinically relevant in the opinion of the investigator
7. Fitzpatrick skin phototype IV-VI
8. Lactating or pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2019-09-02 (Actual); Study Completion 2019-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merete Haedersdal, MD, DMSc, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Department of Dermatology, Bispebjerg Hospital, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Basal Cell Carcinoma Patients
Started | 20
Completed | 19
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Basal Cell Carcinoma Patients
Number analyzed (Participants) | 19
Age, Continuous [Mean (Full Range); unit: years] | 73 [56 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Histological Tumor Subtype [Number; unit: Tumors] — Tumor subtype was determined by pathological analysis of preceding biopsy.
  Tumors
    Nodular BCC | 13
    Superficial BCC | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Occurence of Local Skin Reaction (LSR) Side Effects TOTAL COMPOSITE SCORE
Description: Non-blinded, clinical evaluation of local erythema, edema, flaking, crusting/scabbing, pustulation, scarring, hypo/hyperpigmentation, infection in treated areas will be performed by a physician using a FDA-approved LSR scale at Days 1, 3-5, 14, 30 and 3 months after AFL exposure. Each parameter was graded on a standardized 5-point severity scale (0-4) representing none, mild, moderate, prominent, and severe. A total composite score reflecting overall LSR severity was then calculated based on the sum of all parameters (minimum score 0- least severe; max score: 24-most severe). lower scores are better.
Time Frame: Days 1, 3-5, 14, 30 and 3 months post treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Basal Cell Carcinoma Patients
Number analyzed (Participants) | 19
score on a scale
  Day 1 post treatment | 7 [6 to 9]
  Day 3-5 post treatment | 9 [6 to 11]
  Day 30 post treatment | 4 [2 to 6]
  Month 3 post treatment | 2 [1 to 3]

2. Secondary Outcome: Tumor Response- Clinical Clearance Determined by Clinical Assessment by Physician
Description: Tumor clearance (yes or no) will be evaluated clinically at Day 30 and Month 3. If residual tumor is identified at 3 months follow-up, patients will receive conventional treatment according to national guidelines.¨
Time Frame: Day 30 and Month 3 post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Basal Cell Carcinoma Patients
Number analyzed (Participants) | 19
Participants
  Clinical Clearance Day 30 | 13
  Clinical Clearance Month 3 | 18

3. Secondary Outcome: Imaging-based Tumor Response: Complete Tumor Clearance Determined by Physician Performing Imaging
Description: Clearance (yes or no) will be evaluated using non-invasive dynamic optical coherence tomography, high-intensity focused ultrasound and reflectance confocal microscopy imaging at Day 30 and Month 3. If residual tumor is identified at 3 months follow-up, patients will receive conventional treatment according to national guidelines.
Time Frame: Day 30 and 3 months post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Basal Cell Carcinoma Patients
Number analyzed (Participants) | 19
Participants
  Day 30 | 13
  Month 3 | 18

4. Secondary Outcome: Tumor Response- Histological Tumor Clearance Determined by Pathologist
Description: Histological verification of tumor clearance will be performed 3 months after first treatment using tissue sections from a 4 mm punch biopsy. If residual tumor is identified at 3 months follow-up, patients will receive conventional treatment according to national guidelines.
  NOTE: Overall Number of Participants Analyzed is not consistent with numbers provided in any of the rows in the Participant Flow module since only 18 of the 19 patients consented to undergoing histologicla verification with biopsy. Those, presented data represents patients that underwent biopsy at the 3 month mark.
Time Frame: 3 months post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Basal Cell Carcinoma Patients
Number analyzed (Participants) | 18
Participants | 17

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Basal Cell Carcinoma Patients
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

LIMITATIONS AND CAVEATS:
Readers must be cognizant of the study's unblinded design, lack of conventional treatment control, limited sample size, short follow-up time, and use of punch biopsy rather than excision for histological clearance evaluation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-03): https://cdn.clinicaltrials.gov/large-docs/52/NCT03541252/Prot_SAP_000.pdf